CLINICAL TRIAL: NCT00144027
Title: Patient-Centered Medication Adherence Intervention for Schizophrenia
Acronym: AMAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: IIR 03-257
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Results first posted 2014-12-23 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-07

CONDITIONS: Schizophrenia
Keywords: patient non-adherence; intervention studies
MeSH Terms: conditions — Schizophrenia; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control group will receive treatment as usual; meaning patients in the control group will not receive the medication adherence intervention.
- Antipsychotic adherence intervention (Experimental): Antipsychotic Medication Adherence Intervention which included the Barriers, Facilitators, and Motivators Checklist summary and Adherence tips provided in hard copy to patient and electronic copy to mental health provider.
  Interventions: Behavioral: Antipsychotic medication adherence intervention

INTERVENTIONS:
Behavioral: Antipsychotic medication adherence intervention — The medication adherence intervention will include using a computer to complete a brief set of questions related to medication adherence before mental health clinic visits.
  Arms: Antipsychotic adherence intervention

SUMMARY:
Efficacious antipsychotic medication treatments for schizophrenia are available; however , antipsychotic regimens frequently do not achieve their potential because of poor medication adherence. To date, medication adherence interventions have not been widely adopted or sustained in "real-world" practice settings. One reason for this is the substantial resource investment necessary to implement and sustain available interventions. In response to these problems, we developed a patient-centered adherence intervention based on patient-identified barriers, facilitators, and motivators (BFMs) for medication adherence. The intervention includes a BFM survey (checklist and preference weighting exercise to determine the patient's most important BFM) and a brief list of adherence enhancing suggestions (Options List) tailored to the patient-identified BFMs and compatible with CPRS. The long-term objective of this proposed research is to improve antipsychotic medication adherence and clinical outcomes for patients with schizophrenia using a cost-effective medication adherence intervention. The short-term objectives are to refine and test a patient-centered medication adherence intervention for VA patients with schizophrenia and specifically to: 1. Enhance the feasibility and acceptability of the BFM intervention by reducing the burden on patients and mental health providers through BFM checklist item reduction, provider intervention input, and patient intervention input. We hypothesize that our use of end-user input will result in at least 80% of intervention patients having documentation of a BFM intervention in CPRS. 2. Compare the effects of the BFM intervention versus usual care on changes in medication adherence and schizophrenia symptom severity. We hypothesize that the intervention will result in a) greater medication adherence and b) lower schizophrenia symptom severity than usual care. 3. Exploratory objective: compare the effects of the BFM intervention versus usual care on changes in patient health-related quality of life. We hypothesize that the intervention will result in greater health-related quality of life than usual care.

DETAILED DESCRIPTION:
BFM intervention refinement will be accomplished in five phases. Phase one will include reducing the number of items in the BFM checklist by administering the expanded checklist to at least 50 patients with schizophrenia and using the standard psychometric item-reduction strategies to create a shorter checklist. In phase two we will conduct mental health provider focus groups to discuss the content of the Options List and the delivery of the intervention. In phase three we will automate the BFM intervention using an existing web-based computer touch-screen platform. In phase four we will conduct individual patient debriefing interviews with 30 patients to evaluate the understandability of the BFM survey. In phase five we will evaluate the test/re-test reliability of the survey in a new sample of 30 patients. BFM intervention implementation will include a stratified randomization of patients to the BFM intervention or usual care. BFM intervention evaluation will include testing the feasibility, acceptability, and outcomes associated with the intervention versus usual care in a single trial with 200 patients (100 intervention and 100 usual care).

ELIGIBILITY:
Inclusion Criteria:

* medical chart diagnosis of schizophrenia or schizoaffective disorder;
* currently prescribed outpatient antipsychotic medication (oral or depot);
* patient must have adequate capacity to provide informed consent, understand the nature of the study, and sign an informed consent document.

Exclusion Criteria:

- significant cognitive impairment as indicated by a score > 10 on the Blessed Orientation-Memory-Concentration (BOMC) Test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-12; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Pyne, MD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas, United States

REFERENCES:
- [Result] Pyne JM, Fischer EP, Gilmore L, McSweeney JC, Stewart KE, Mittal D, Bost JE, Valenstein M. Development of a Patient-Centered Antipsychotic Medication Adherence Intervention. Health Educ Behav. 2014 Jun;41(3):315-24. doi: 10.1177/1090198113515241. Epub 2013 Dec 25. PMID 24369177

RESULTS

PARTICIPANT FLOW:
Groups:
- Antipsychotic Adherence Intervention Group: Antipsychotic medication adherence intervention: The medication adherence intervention will include using a computer to complete a brief set of questions related to medication adherence before mental health clinic visits. The patient will receive a hard copy summary of their responses (top 3 barriers and top 3 facilitators and motivators) with brief adherence tips which are specific to the patient-selected barriers. The provider will received the same information in an electronic health record adherence note.
Period: Overall Study
Arm/Group | Control | Antipsychotic Adherence Intervention Group
Started | 39 (participants who consented) | 36 (participants who consented)
Completed Baseline Assessment | 39 | 29
Completed 6 Month Assessment | 37 | 24
Completed | 36 (participants who completed 12-month follow-up) | 25 (participants who completed 12-month follow-up)
Not Completed | 3 | 11
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — did not complete baseline assessment | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Control/No Intervention: The control group will receive treatment as usual; meaning patients in the control group will not receive the medication adherence intervention.
- Intervention Group: Antipsychotic medication adherence intervention: The medication adherence intervention will include using a computer to complete a brief set of questions related to medication adherence before mental health clinic visits. The patient will receive a hard copy summary of their responses (top 3 barriers and top 3 facilitators and motivators) with brief adherence tips which are specific to the patient-selected barriers. The provider will received the same information in an electronic health record adherence note.
- Total: Total of all reporting groups
Arm/Group | Control/No Intervention | Intervention Group | Total
Number analyzed (Participants) | 39 | 29 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (8.3) | 52.9 (5.6) | 53.3 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 36 | 25 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 22 | 45
  White | 16 | 7 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Antipsychotic Medication Adherence
Description: The self-report adherence measure asked patients to think about the past four weeks and report to what extent they took their medication for mental, emotional, or nervous problems and report the result on a 5-point Likert scale ranging from 'I never missed taking my medicine' to 'I stopped taking the medicine altogether'. Patients who received depot injections were asked to think about the past six months. Self-report adherence was defined as 1=I never missed taking my medicine' and 0=any other response to the medication adherence question.
Time Frame: 6-months
Population: Percent of participants who reported "never missed taking my medication" at 6-months
Measure: Number; unit: percentage of participants
Arm/Group | Control/No Intervention | Intervention Group
Number analyzed (Participants) | 37 | 24
percentage of participants | 63.9 | 75.0
Statistical Analysis 1: Comparison: Control/No Intervention vs Intervention Group; Test type: Superiority or Other; p = 0.03, Regression, Logistic; logistic regression predicting 6-month adherence, controling for baseline depression, extrapyramidal side effects, and baseline adherence; Odds Ratio (OR) = 7.57, 95% CI 2-sided [1.21 to 47.53]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control/No Intervention | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/30
Other Adverse Events (participants affected / at risk) | 0/39 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes